CLINICAL TRIAL: NCT03338374
Title: Heart Failure With Preserved Ejection Fraction Treated by Cardiac Resynchronisation Therapy Versus Rate Responsive Pacing: A Mechanistic Study
Brief Title: Cardiac Resynchronisation Therapy Versus Rate-responsive Pacing in Heart Failure With Preserved Ejection Fraction
Acronym: PREFECTUS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cardiff and Vale University Health Board (Other Government)
Collaborators: Abbott (Industry); Cardiff Metropolitan University (Other)
Responsible Party: Principal Investigator, Freya Lodge, Clinical Research Fellow, Cardiff and Vale University Health Board
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17/WA/0004 190938
Record Dates: First submitted 2017-08-31; First posted 2017-11-09 (Actual); Last update posted 2023-06-02 (Actual); Status verified 2023-06

CONDITIONS: Diastolic Heart Failure
Keywords: Cardiac chronotropy; Cardiac resynchronisation therapy; Rate responsive pacemaker; Heart failure with preserved ejection fraction
MeSH Terms: conditions — Heart Failure, Diastolic | interventions — Cardiac Resynchronization Therapy Devices

STUDY DESIGN:
Intervention Model Description: Exploratory single-centre, open label, non-randomised, prospective cohort study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Biventricular Pacemaker (Experimental): All subjects to be in a single study group experiencing all interventions.
  Interventions: Device: Biventricular pacemaker

INTERVENTIONS:
Device: Biventricular pacemaker — All subjects will receive a biventricular pacemaker at implantation. Programming will initially be to dual-chamber, dual-function rate-responsive pacing for 12 weeks; following reassessment, device will be reprogrammed to biventricular pacing for a further 12 weeks. Optional study extension: if incremental benefit is shown for biventricular pacing above dual chamber, the mechanism will be sought using echocardiographic evidence and the devices will be optimised according to this mechanism of action to see whether further benefit can be achieved.
  Other Names: Rate responsive pacing

SUMMARY:
Half of patients with heart failure have normal heart pumping function (Heart failure with Preserved Ejection Fraction, HFpEF), most commonly characterised by breathlessness on exercise. A number of mechanisms are responsible, but frequently patients are unable to raise their heart rate on exercise. This can be treated by a 'rate-responsive pacemaker' (RRP), which detects exercise and increases the heart rate accordingly. Some beneficial effects on echocardiographic parameters have been reported with exercise programmes. However, evidence based treatment options are limited in this group and therapy mainly relies on water tablets and treatment of blood pressure.

Cardiac resynchronisation therapy (CRT) is a technique using specialised 'biventricular' pacemakers that is well established in heart failure with reduced pump function. Patients who respond to this treatment have lower risk of death and hospitalisation and usually feel better. CRT is not currently used in HFpEF. The PROSPECT trial showed that some patients with relatively preserved heart function exhibited similar benefits to those with poor pump function, but this has not been formally tested. CRT aims to make the heart beat in a more synchronised way. Patients with HFpEF commonly have evidence of reduced heart synchronisation.

The investigators plan to assess the feasibility of using a prospective cohort study to assess the incremental benefit of CRT over and above RRP in patients with HFpEF. 10 patients with HFpEF and insufficient heart rate will be recruited and will undergo exercise testing, heart scanning and symptom questionnaires. A biventricular pacemaker will be implanted and programmed to RRP for 12 weeks before repeating the tests. After this, the investigators will non-invasively programme the pacemaker to CRT for 12 weeks and repeat the functional tests. If incremental benefit is shown with CRT the echocardiograms will be analysed in detail to determine the mechanism of change. The study participants will be invited to continue their involvement in a study extension. This will involve non-invasively programming the pacemakers to optimise their function guided by the results of the echocardiograms in the first two phases of the study. After a further 12 weeks, the functional assessments will be repeated. If no benefit is seen with CRT after initial analysis, the participant involvement will end.

DETAILED DESCRIPTION:
This is an exploratory single-centre, open label, non-randomised, prospective cohort study comparing rate responsive pacing (RRP) with CRT in patients with confirmed HFpEF and chronotropic incompetence.

Setting:

The study will be conducted in Cardiff and Vale University Health Board, with patients drawn from Cardiology clinics and inpatient wards. Follow-up assessments will be conducted at Cardiff School of Sport, a research facility at a university campus close to the main hospital.

Number of subjects planned:

10 patients. This will be sufficient to establish estimates of variability in the diastolic reserve index (see below), allow estimation of treatment difference and gauge acceptability.

Target population:

Subjects with HFpEF and chronotropic incompetence

Endpoints:

Systolic and diastolic longitudinal reserve index are calculated by the following formulae:

Systolic reserve = Δs' x [1-(1/s'rest)] Diastolic reserve = Δe' x [1-(1/e'rest)]

These are known to be impaired in patients with HFpEF and are a marker of adaptation to exercise in terms of filling pressures and left ventricular relaxation. Tan et al report a significant difference between the results seen with 56 patients with HFpEF and 27 control subjects on exercise echocardiography with semi-supine bicycle.16 Patient characteristics were similar to those of our proposed study group (Ejection fraction (EF) >50%, New York Heart Association (NYHA) classification grade II, HFpEF according to Vasan and Levy criteria).28

The investigators will therefore investigate diastolic and systolic reserve index as possible endpoints of a future study into the efficacy of CRT versus RRP in HFpEF patients.

Planned interventions:

Visit 1 - Baseline Assessments: Patients will undergo initial assessment of baseline characteristics by echocardiography, cardiopulmonary exercise testing, 6-minute walk test (6MWT) and Minnesota Living with Heart Failure Questionnaire (MLHFQ). (Visit length: approx. 4 hours)

Visit 2 - Device Implantation (≤ 7 days after baseline assessments completed):

Eligible subjects will undergo implantation of a biventricular pacemaker under normal laboratory conditions. The device will be programme to administer rate-responsive pacing (DDDR). They will return to pacing clinic a week later for a programming check; during this visit, they will also undergo a chest x-ray according to local protocol to ensure correct lead placement (Visit length: 1 day + 2 hours)

Visit 3 - Assessments and Device Reprogramming After 12 weeks, the baseline parameters will be reassessed and patients will then have their device non-invasively reprogrammed to CRT. (Visit length: approx. 4 hours)

Visit 4 - Assessments After a further 12 weeks, the baseline assessments will be repeated. The pacemaker will be non-invasively reprogrammed to DDDR mode and the patient will go home. (Visit length: approx. 4 hours)

Optional extension (pending analysis of results) Visit 5 - Reprogramming If incremental benefit has been demonstrated with CRT above the benefit of RRP, the echocardiograms will be examined to establish the mechanism of improvement. Subjects will be invited to participate in a study extension using multisite technology. The device will be non-invasively reprogrammed to optimise the CRT settings targeted specifically for the mechanism identified. (Visit length: approx. 3 hour)

Visit 6 - Assessments 12 weeks after the final reprogramming, patients will attend for a final set of assessments as per baseline. Participant involvement will then cease. (Visit length: approx. 4 hours)

Total contact time with research team: Approximately 27 hours (22 hours without extension)

ELIGIBILITY:
Inclusion Criteria:

* Confirmed HFpEF as described above
* Chronotropic incompetence as described above
* Ongoing exertional breathlessness of NYHA Grade II or worse
* Ability to understand and sign written consent form
* Males and females, age >18 years
* Ability to participate in follow-up appointments at 3 and 6 months post-implantation
* Ability to complete a cardiopulmonary exercise test

Exclusion Criteria:

* Any contraindication to implantation of permanent pacemaker, namely unresolved infective process or sepsis, vascular access difficulties, advanced neoplastic process, expected lifespan less than 1 year or patient choice
* Ejection fraction <50%
* Known valvular disease graded severe or moderate-to-severe
* Cardiac arrhythmia (paroxysmal or persistent) within 1 year of recruitment
* Exertional chest pain suggestive of angina or personal history of coronary artery disease without subsequent revascularisation, or coronary angiogram within the past 5 years demonstrating >50% stenosis in ≥ 1 epicardial coronary artery
* Significant chronic lung disease (FEV1 <80%)
* Inability to complete follow-up process for any reason not defined above

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-11-27 (Actual); Primary Completion 2022-05-30 (Actual); Study Completion 2022-05-30 (Actual)

PRIMARY OUTCOMES:
Diastolic reserve index | After 12 weeks of rate responsive pacing and again after 12 weeks of biventricular pacing; study extension: after 6 weeks of optimised pacing
  The change in e' between rest and exercise, as measured by tissue Doppler in the septal and/or lateral left ventricular walls on echocardiography. To be expressed using the formula: [change in e'] x [1-(1/e' at rest)]. e' is the peak diastolic velocity of the myocardium during passive left ventricular filling.
Systolic reserve index | After 12 weeks of rate responsive pacing and again after 12 weeks of biventricular pacing; study extension: after 6 weeks of optimised pacing
  The change in s' between rest and exercise, as measured by tissue Doppler in the septal and/or lateral left ventricular walls on echocardiography. To be expressed using the formula: [change in s'] x [1-(1/s' at rest)]. s' is the peak systolic velocity of the myocardium.

SECONDARY OUTCOMES:
Global longitudinal strain | After 12 weeks of rate responsive pacing and again after 12 weeks of biventricular pacing; study extension: after 6 weeks of optimised pacing
  Peak systolic strain of 6 myocardial segments measured on echocardiography by speckle tracking, measured both at rest and on exercise
Left ventricular torsion | After 12 weeks of rate responsive pacing and again after 12 weeks of biventricular pacing; study extension: after 6 weeks of optimised pacing
  The twisting movement of the heart can be quantified with echocardiography using speckle tracking at rest and on exercise.
Exercise duration | After 12 weeks of rate responsive pacing and again after 12 weeks of biventricular pacing; study extension: after 6 weeks of optimised pacing
  Cardiopulmonary exercise testing will be used with standard local protocols to evaluate exercise duration.
Oxygen carrying capacity | After 12 weeks of rate responsive pacing and again after 12 weeks of biventricular pacing; study extension: after 6 weeks of optimised pacing
  Measurement of peak ventilatory capacity (VO2 max) using cardiopulmonary exercise testing with standard local protocols, ensuring a respiratory exchange ratio of greater than 1.1 to guarantee near-maximal exercise achieved. This will be assessed using expired gas analysis, which is a standard technique.
Distance walked in a six-minute walk test | After 12 weeks of rate responsive pacing and again after 12 weeks of biventricular pacing; study extension: after 6 weeks of optimised pacing
  Subjects walk down a pre-measured course, usually a hallway or corridor, and their distance achieved after six minutes is recorded.
New York Heart Association Function Class | After 12 weeks of rate responsive pacing and again after 12 weeks of biventricular pacing; study extension: after 6 weeks of optimised pacing
  Standard measure of heart failure severity that correlates with outcomes. Assessed using measures of impairment in activities of daily living, such as dressing, walking.
Minnesota Living with Heart Failure Quality of Life Score | After 12 weeks of rate responsive pacing and again after 12 weeks of biventricular pacing; study extension: after 6 weeks of optimised pacing
  Change in Minnesota living with heart failure questionnaire score. This questionnaire asks 21 questions relating to daily tasks of living, hobbies, social life and well-being in relation to heart failure symptoms and ascribes greater points to more severe symptoms; a higher score is therefore indicative of a lower quality of life. Scores may range between 0 and 105.
Prognostic biomarkers | After 12 weeks of rate responsive pacing and again after 12 weeks of biventricular pacing; study extension: after 6 weeks of optimised pacing
  Measurement of serum N-terminal pro-B-type Natriuretic Peptide, a commonly used marker of ventricular wall stretch that correlates with heart failure severity and is adversely associated with prognosis.

OTHER OUTCOMES:
Drop-out rate | At 24 weeks (or if study extension used, then following completion of this 6-week extension)
  A measure of the number of participants who fail to complete the study processes, to inform further studies using a similar design

CONTACTS AND LOCATIONS:
Overall Officials: Zaheer Yousef, MD, Study Director — Cardiff and Vale University Health Board
Locations (2):
- United Kingdom (2):
  - Cardiff and Vale University Health Board, Cardiff, Mid Glamorgan
  - Cardiff Metropolitan University, Cardiff, Mid Glamorgan

IPD SHARING:
Plan to Share IPD: No
Access to individual participant data (IPD) will be at the discretion of the study team. No plan is currently in place to share IPD. This is a small, exploratory study where full transparency will be demonstrated in publication of results; fully-anonymised individual participant data may be referenced in publication of results.

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-09-14): https://cdn.clinicaltrials.gov/large-docs/74/NCT03338374/Prot_SAP_001.pdf
  • Informed Consent Form (2017-05-15): https://cdn.clinicaltrials.gov/large-docs/74/NCT03338374/ICF_000.pdf